CLINICAL TRIAL: NCT00439348
Title: Improving Over-the-counter Medication Compliance.
Brief Title: Over-the-Counter Medication Usage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: D. Ashley Hill, M.D., Florida Hospital Department of Obstetrics and Gynecology
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 07.02.01
Record Dates: First submitted 2007-02-21; First posted 2007-02-23 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Drugs, Non-Prescription; Medication Systems
Keywords: Calcium; Compliance; Medication compliance; electronic prescription; over-the-counter medications; OTC medications
MeSH Terms: conditions — Patient Compliance; Medication Adherence | interventions — Prescriptions

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Electronic prescription (Experimental): Patients receive a prescription for specific over-the-counter medications.
  Interventions: Behavioral: Prescription
- Verbal advice (Active Comparator)
  Interventions: Behavioral: Verbal advice

INTERVENTIONS:
Behavioral: Verbal advice — Patients receive verbal advice regarding specific over-the-counter medications.
  Arms: Verbal advice
Behavioral: Prescription — Patients receive a prescription for a specific over-the-counter medication.
  Arms: Electronic prescription

SUMMARY:
There are several benefits of over-the-counter medications, yet there is little research evaluating how to increase patient compliance when a health care provider suggests an over-the-counter (OTC) medication. We are evaluating two types of physician directions to see which increases patient compliance with OTC medications.

DETAILED DESCRIPTION:
Researchers will identify a cohort of gynecologic patients presenting for annual examinations and offer participation in the study. Physician researchers will randomize patients to 2 types of physician directions about OTC medications, then follow compliance over the course of the next 7 months. A total of 123 participants in each arm will undergo recruitment, until a total of 246 participants are recruited.

Inclusion criteria include: female, non-pregnant patients presenting for annual gynecologic examinations between the ages of 19-50.

Exclusion criteria include: outside of study age range, patient taking thyroid medication, history of kidney stones, history of hypercalcemia, non-English speaking.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing annual gynecologic examinations.
* Ages 19-50.
* Patients not currently taking certain OTC medications.

Exclusion Criteria:

* Pregnancy.
* History of hypercalcemia.
* History of kidney stones.
* Outside study age range of 19-50.
* Patient taking thyroid medication.

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 246 (Actual)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Determining which of 2 types of physician direction regarding OTC medication usage improves patients compliance, as assessed at 3 and 6 months after enrollment. | 3 and 6 months after enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: D. A Hill, MD, Study Chair — Department of Obstetrics and Gynecology, Florida Hospital Family Medicine Residency Program
Locations (1):
- Loch Haven Ob/Gyn Group, Orlando, Florida, United States